CLINICAL TRIAL: NCT01906424
Title: Restoring Arm and Hand Function With Non-invasive Spinal Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NeuroEnabling Technologies, Inc. (Industry)
Collaborators: University of California, Los Angeles (Other); California Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: NETI201307
Record Dates: First submitted 2013-07-16; First posted 2013-07-24 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2016-04

CONDITIONS: Paralysis; Spinal Cord Injury
Keywords: spinal cord injury; quadriplegia; tetraplegia; stimulation
MeSH Terms: conditions — Paralysis; Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control Grp#1: Training w/ and w/o Stim (Other): Control- Group #1: 4 weeks training without any transcutaneous electrical stimulation followed by 2 weeks of training plus transcutaneous electrical spinal cord stimulation applied to one or two locations of the cervical (neck) region of the spinal cord.
  Interventions: Device: Transcutaneous Electrical Spinal Cord Stimulation
- Grp#2: Training+Single Site Stimulation (Active Comparator): Group #2: Four weeks of training plus transcutaneous electrical spinal cord stimulation applied to one location along the cervical (neck) region of the spinal cord; followed by 2 weeks of training without stimulation
  Interventions: Device: Transcutaneous Electrical Spinal Cord Stimulation
- Grp #3: Training + Two Site Stimualtion (Active Comparator): Group #3: Four weeks of training plus transcutaneous electrical spinal cord stimulation applied to two locations along the cervical (neck) region of the spinal cord; followed by 2 weeks of training without stimulation
  Interventions: Device: Transcutaneous Electrical Spinal Cord Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Spinal Cord Stimulation — A prototype device that delivers transcutaneous electrical stimulation will be used to stimulate the cervical spinal cord.
  Other Names: Prototype device

SUMMARY:
This study is to determine if non-invasive electrical stimulation of the spinal cord can help improve hand and arm function in people with paralysis who suffered a cervical spinal cord injury.

DETAILED DESCRIPTION:
This study is to determine if non-invasive electrical stimulation of the spinal cord can help improve hand and arm function in people with paralysis who suffered a cervical spinal cord injury. The investigators hypothesize that this stimulation can revive spared function in the spinal cord of individuals who are clinically paralyzed, but who have some remaining connections between the brain and spinal cord. Our research has demonstrated that modifying the activation state of the spinal cord or awakening the spinal cord can benefit people with paralysis years after a spinal cord injury. This method and device have not yet been approved by the FDA for the treatment of paralysis and are under investigation. This study if successful will help provide further evidence that could be use to gain FDA approval.

ELIGIBILITY:
Inclusion Criteria: ASIA C

* Spinal cord injury 1 or more years prior
* Non progressive SCI at C7 or higher
* Half of key muscles below neurological level having a motor score of less than 2/5
* Ability to commit to home exercises and 12 week participation
* Stable medical condition without cardiopulmonary disease or dysautonomia that would contraindicate participation in upper extremity rehabilitation or testing activities
* Not dependent on ventilation support
* No painful musculoskeletal dysfunction, unhealed fracture, pressure sore, or urinary tract infection that might interfere with upper extremity rehabilitation or testing activities
* No clinically significant depression or ongoing drug abuse
* Adequate social support network to be able to participate in weekly training and assessment sessions for the duration of the 12 week study period
* No current anti-spasticity regimen
* Must not have received botox injections in the prior six months
* Be unable to use upper extremity for functional tasks

Exclusion Criteria:

* Pregnancy
* No functional segmental reflexes below the lesion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-04; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement in sensorimotor function in arms and hands | 12 weeks
  Subjects will be tested by several measures of sensory and motor function, as well as self-assessments regarding quality of life and independence, at the beginning of the study and at each testing session. These tests include:
  American Spinal Injury Association (ASIA) scoring system. Box and block CUE (Capabilities of Upper Extremity) GRASSP (Graded Redefined Assessment of Strength, Sensibility and Prehension) SCIM (Spinal Cord Independence Measure)
  Ashworth Spasticity scale:
  Penn Spasm Frequency VAS (Visual Analog Scale) for Spasticity)

CONTACTS AND LOCATIONS:
Overall Officials: Victor R Edgerton, PhD, Study Chair — University of California, Los Angeles; Nicholas Terrafranca, DPM, Principal Investigator — NeuroEnabling Technologies, Inc.
Locations (2):
- United States (2):
  - University of California Los Angeles, Los Angeles, California
  - Strides SCI Functional Fitness, San Juan Capistrano, California